CLINICAL TRIAL: NCT07033871
Title: Comprehensive Geriatric Assessment in Chronic Disease Management for Older Adults in China: A Registry Study （CGACDM - Older Adults in China）
Acronym: CGACDM - Older
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Provincial People's Hospital (Other)
Collaborators: Geriatrics Research Institute of Henan Provincial People's Hospital (Unknown); Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: HenanPPH-CGA
Record Dates: First submitted 2025-05-26; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-05

CONDITIONS: Comprehensive Geriatric Assessment; Chronic Disease Management; Older Adults (65 Years and Older)
Keywords: Comprehensive Geriatric Assessment; Chronic Disease Management; Older Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elderly patients with chronic diseases: The study population consisted of patients with chronic diseases in the elderly who underwent comprehensive geriatric assessment and management. Chronic diseases in the elderly included but were not limited to chronic heart failure, chronic obstructive pulmonary disease, cognitive dysfunction, and so on. We compared various biochemical indexes, cardiac function indexes, quality of life, and the occurrence of long-term adverse events before and after the comprehensive geriatric assessment and management.
  Interventions: Diagnostic Test: comprehensive geriatric assessment
- Healthy elderly population: The control group was composed of elderly subjects without evidence of chronic diseases. Chronic diseases was excluded by performing a complete medical history, a comprehensive physical examination, and an echocardiogram.
  Interventions: Diagnostic Test: comprehensive geriatric assessment

INTERVENTIONS:
Diagnostic Test: comprehensive geriatric assessment — The comprehensive geriatric assessment (CGA) is a multi dimensional diagnostic process used to determine the medi cal, psychological, and functional capabilities of a frail elderly person to develop a coordinated and integrated plan for treat ment and long-term follow-up.

SUMMARY:
With the continuous development of China's economy and the improvement of medical standards, the life expectancy of the Chinese population has significantly increased. Against the backdrop of accelerating aging in China, the incidence of age-related chronic non-communicable diseases (NCDs), such as cardiovascular and cerebrovascular diseases and chronic respiratory diseases, has risen remarkably. These diseases are characterized by multiple comorbidities, high disability rates, and high mortality rates, severely compromising the quality of life of older adults, exacerbating family burdens, and straining healthcare systems. This constitutes one of the major challenges faced by aging societies. Therefore, early detection and intervention of chronic diseases in older adults are critical measures to address population aging.

Comprehensive geriatric assessment (CGA), a core specialty of geriatric medicine, serves as a fundamental framework for the clinical identification of geriatric syndromes and multidisciplinary management. It is emerging as a key pathway to promote "healthy aging." Guided by this premise, this study aims to explore the application value of CGA in managing chronic diseases among older adults, with the goal of achieving full-cycle management for early detection, diagnosis, and treatment of chronic conditions in China's elderly population.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 60 years or older 2. Diagnosed with chronic diseases in the circulatory, respiratory, digestive, nervous, or endocrine systems, consistent with corresponding disease diagnostic criteria; 3. Availability of complete medical records; 4. Clear consciousness and ability to independently answer questions; 5. Signed informed consent form.

Exclusion Criteria:

* 1. Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient (e.g. tourist, non-native speaker or does not understand the local language, psychiatric disturbances).

  2. Presence of serious/severe co-morbidities in the opinion of the investigator which may limit short term (i.e. 6 month) life expectancy.

  3. Current participation in a randomised interventional clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients with chronic diseases in the elderly who underwent comprehensive geriatric assessment and management. Chronic diseases in the elderly included but were not limited to chronic heart failure, chronic obstructive pulmonary disease, cognitive dysfunction, and so on.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Major adverse events (MAE) | These data is collected during follow-up visit at 3/6/12/24/36 months after discharge
  Major adverse events (MAE) in overall population, defined as composite of all-cause death, Heart Failure hospitalization, recurrent myocardial infarction, stroke, etc.

OTHER OUTCOMES:
Age for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Gender for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Height for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Weight for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Contact information for each participant | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Past Medical History including disease history, surgical history, and family medical history | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Lifestyle including smoking history and drinking, specify how many years smoking or drinking lasted and detail quantity per day | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：blood lipid | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：blood glucose | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：uric acid | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：urea | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：creatinine | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：C reactive protein | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：D-dimer | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
blood biochemical index：NT-proBNP | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
Cardiac ultrasound | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  The whole results of echocardiography report will be recorded. The indicates which can reflect cardiac function including Left ventricular ejection fraction, left ventricular end diastolic diameter, E/A ratio of bicuspid valve will be used to calculate the association with metabolites.
Drug treatment | These data is collected from the cases' medical record in an average of 1 month after the sample recruiting
  Oral drug therapy, including antiplatelet drugs, antihypertensive drugs, lipid-lowering drugs, etc.
Comprehensive Geriatric Assessment: Frailty | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Sarcopenia | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Falls | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Disability | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Dysphagia | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Malnutrition | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Urinary incontinence | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Fecal incontinence | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Constipation | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Cognitive impairment | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Anxiety state | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Depressive state | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Sleep disorders | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Pain | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Social support | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment
Comprehensive Geriatric Assessment: Home environment | These data were collected from the comprehensive geriatric assessment process within an average of 1 week after sample recruitment

IPD SHARING:
Plan to Share IPD: No